CLINICAL TRIAL: NCT02995200
Title: Quantification of Upper Extremity Use and Effects of Feedback in the Home Setting
Acronym: UnSumRes2015
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland State University (Other)
Responsible Party: Principal Investigator, Maureen Whitford, Assistant Professor, Cleveland State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2016-182
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Feedback Intervention (Participants Post-stroke); Healthy Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Post-Stroke (Experimental): 2 sessions of in-home accelerometer based feedback about paretic arm use
  Interventions: Behavioral: Accelerometer Based Feedback
- Healthy Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Accelerometer Based Feedback
  Arms: Group Post-Stroke

SUMMARY:
A pilot study, the purpose of which is to use accelerometers to quantify UE use (1 and two hand use) in healthy controls and people post-stroke from which the investigators will develop use-based feedback to improve recovery in the home setting. The objectives of this pilot study are to:

i.) determine the feasibility of using accelerometers to quantify amount of UE use in the home setting in healthy individuals and individuals chronic post-stroke,

ii.) quantify and compare the unilateral activity of the weaker (paretic) versus stronger (non-paretic) UEs,

iii.) quantify and compare amount of UE use in healthy controls to that of people chronic post-stroke (side matched unimanual use for each arm and bilateral use) in the home, and

iv.) assess the effect of a few sessions of in-home accelerometer used-based feedback on unilateral and bilateral UE use.

v.) assess kinematic, kinetic, and EMG data during UE movements bilaterally and between healthy controls and subjects post-chronic stroke pre and post feedback (for the people after stroke).

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adults: 40-100 years old, able to follow 2-step commands, able to comply with experimental protocol, living in a home setting, full active range of motion (AROM) in both shoulders and elbows for their age group.
* Individuals Post-stroke: Able to follow 2-step commands, 40 - 100 years old, community dwelling with or without assistance, no upper extremity (UE) injury within the last 3 months, at least 30 degrees of flexion AROM (with or without assistance) and PROM in shoulder and elbow in or out of synergy, intact superficial light touch sensation in both UEs, and at least 6 months post ischemic or hemorrhagic stroke that is either cortical, subcortical or in the cerebellum. It does not need to be their first and only stroke.

Exclusion Criteria:

* Healthy Adults: Injury of either UE within the last 3 months and unable to follow commands related to the accelerometer use/protocol.
* Individuals Post-stroke: Unable to follow 2 step commands, inability to adhere to study requirements, any neurological diagnosis other than stroke (i.e. Parkinson's Disease, Multiple Sclerosis, etc.), and aphasia limiting their ability to complete the MoCA and Stroke Impact Scale (SIS) questions.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Amount of Use (measured by accelerometer) | 3 week period

IPD SHARING:
Plan to Share IPD: No